CLINICAL TRIAL: NCT04093804
Title: Impact of Glenosphere Size on Range of Motion in Female Patients Undergoing Reverse Shoulder Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondren Orthopedic Group L.L.P. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOH183
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Rotator Cuff Tear Arthropathy; Massive Irreparable Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Intervention Model Description: This study is a randomized trial consisting of female patients undergoing reverse shoulder arthroplasty for rotator cuff tear arthropathy or a massive irreparable rotator cuff tear. The experimental group will receive a 36mm glenosphere and the control group will receive the standard 32mm glenosphere. All other conditions of the surgical procedure will be identical as well as the clinical follow-up.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 32mm Glenosphere (Active Comparator): The control group will receive the standard 32mm glenosphere.
  Interventions: Device: Glenosphere size for Reverse Shoulder Arthroplasty
- 36mm Glenosphere (Experimental): The experimental group will receive a 36mm glenosphere.
  Interventions: Device: Glenosphere size for Reverse Shoulder Arthroplasty

INTERVENTIONS:
Device: Glenosphere size for Reverse Shoulder Arthroplasty — Two randomized study groups will be formed with the consented patients (experimental and control). All patients will undergo reverse shoulder arthroplasty by the Principal Investigator. The experimental group patients will receive a 36mm glenosphere and the control group will receive a 32mm glenosphere. All other procedures during the surgery are identical between groups.

SUMMARY:
The purpose of this study is to perform a prospective randomized trial among female patients undergoing reverse shoulder arthroplasty (RSA) to determine if a larger glenosphere allows greater range of motion without an impact on complications.

DETAILED DESCRIPTION:
A current research debate is whether glenosphere size has a significant clinical impact on a patient's range of motion (ROM) following RSA. Some researchers have shown an association between increased glenosphere size and improved ROM, but no study has determined the absolute minimal motion differences that would be recognizable or beneficial by patients. This is mostly attributable to limitations such as small sample sizes as well as the fact that shoulder dynamics are multifactorial in nature. Most studies have shown an increased ROM with larger glenosphere sizes.1 Because smaller patients are often times female and receive smaller implants, female patients may be more susceptible to limited ROM. The purpose of this study is to determine if a larger glenosphere allows for greater ROM in female patients undergoing RSA.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Diagnosis of rotator cuff tear arthropathy or a massive irreparable rotator cuff tear for which the patient has elected to undergo reverse shoulder arthroplasty
* No history of prior shoulder arthroplasty
* Consent to study participation by signing the informed consent and the Protected Health Information (PHI) form (Attachment B and C)
* Ability to speak, read and write English

Exclusion Criteria:

* Male sex
* Any impairment that would prevent answering the surveys
* No children or adolescents under the age of 18 years old
* No prisoners, pregnant women, or mentally disabled persons
* No Workers' Compensation cases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Active range of motion | Change from baseline (pre-operative) to 2 years follow-up
  Shoulder elevation, abduction, external rotation in abduction, and internal rotation
Passive range of motion | Change from baseline (pre-operative) to 2 years follow-up
  Shoulder elevation and external rotation

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeon (ASES) Shoulder Index | Change from baseline (pre-operative) to 2 years follow-up
  Standard functional outcomes questionnaire following shoulder surgery, range 0 - 100 (highest function)
Constant-Murley Shoulder Outcome score | Change from baseline (pre-operative) to 2 years follow-up
  Standard functional outcomes questionnaire following shoulder surgery, range 0 - 100 (highest function)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondren Orthopedic Group, L.L.P., Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mollon B, Mahure SA, Roche CP, Zuckerman JD. Impact of glenosphere size on clinical outcomes after reverse total shoulder arthroplasty: an analysis of 297 shoulders. J Shoulder Elbow Surg. 2016 May;25(5):763-71. doi: 10.1016/j.jse.2015.10.027. Epub 2016 Feb 4. PMID 26853756